CLINICAL TRIAL: NCT01246219
Title: The Influence of Growth Hormone (GH) Therapy on Short Stature Related Distress a Prospective Randomized Controlled Trial
Brief Title: Short Stature Related Distress
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: rmc004981ctil
Record Dates: First submitted 2010-11-16; First posted 2010-11-23 (Estimated); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Idiopathic Short Stature; Self Image
Keywords: Idiopathic Short stature; Self Image; GH therapy; Psychological distress
MeSH Terms: interventions — Human Growth Hormone; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- GH treatment (Experimental): 4 years of GH treatment
  Interventions: Drug: GH treatment (Genotropin)
- Placebo (Placebo Comparator): 1 year treatment with placebo followed by optional 3 years of GH treatment
  Interventions: Drug: 1 year treatment with placebo followed by optional 3 years of GH treatment
- Non treatment group (No Intervention)

INTERVENTIONS:
Drug: GH treatment (Genotropin) — 4 years treatment with GH
  Arms: GH treatment
Drug: 1 year treatment with placebo followed by optional 3 years of GH treatment — 1 year treatment with placebo followed by optional 3 years of GH treatment
  Arms: Placebo

SUMMARY:
The research aims to provide data on gender-related psychological impact of GH (Growth Hormone)treatment. Implicit measurable psychological metrics of the therapy outcome on males are to be evaluated in a Prospective Randomized Controlled Trial. As a secondary axis of the study, the investigators aim to provide descriptive documentation of the unique distress signal manifestation implicitly shown by Idiopathic Short Stature (ISS) boys and suggest methods of early detection and measurement of such manifestations that can be used to cement guidelines for the treatment in GH.

DETAILED DESCRIPTION:
Study Design:

A prospective randomized, double blind, placebo controlled trial design, comparing four research groups, with 4 repeated psychological measures (before treatment, after 3 months,after 1 year, and at the end of treatment, after 4 years).

The study will be divided into two segments:

Segment 1:double blind, placebo controlled, will include the first 60 ISS (Idiopathic Short Stature)recruited patients. Patients in this segment will be randomized to one of the growth hormone treatment groups in a ratio of 2:1. 40 patients will be treated 4 years with GH and 20 patients will be treated with placebo at the first year of the study and will have the option to start GH treatment after one year, for a duration of 3 years.

Segment 2:after the enrollment to segment 1 will end, enrollment to segment 2 will begin.Participants in segment 2 (patients with ISS and short stature) will serve as control groups and therefore will not be treated with growth hormone. Patients in Segment 2 will be evaluated only once.

The 4 repeated psychological evaluations (before treatment,after 3 months, after 1 year, and at the end of treatment, after 4 years)will include the following:

1. Implicit Association Test
2. Masculine Self Image
3. Pictures Projective Test
4. The Rosenberg Self Esteem Scale-a self report measure of explicit self- esteem
5. Quality of Life Questionnaire
6. Silhouette Apperception Technique (SAT)- a self report measure assessing children's and adolescent's perception of their own body size compared with that of their age-related peers
7. Child Behavior Checklist

ELIGIBILITY:
Inclusion Criteria:

1 Segment 1 :Boys at the age range of 8-13 years 2. Segment 2: Boys at the age range of 12-17 years 3. Tanner stage 1 (segment 1 only) 4. more than 2 SD's (standard deviation) below the average height

Exclusion Criteria:

1. Mental retardation,
2. Psychiatric illness,
3. Lack of informed consent\assent.
4. Health status that required chronic treatment with steroids

Ages: 8 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Psychological Distress score | After 4 years of treatment
  short stature related distress score as measured by the Height Perception Pictures Test
Psychological Distress score | After 4 years of treatment
  short stature related distress score as measured by the Rosenberg Self-Esteem Scale
Psychological Distress score | After 4 years of treatment
  short stature related distress score as measured by the Quality of Life questionnaire
Psychological Distress score | After 4 years of treatment
  short stature related distress score as measured by Silhouette Apperception Technique questionnaire

SECONDARY OUTCOMES:
Perceived self image score | After 4 years of treatment
  Perceived self image score as measured through Single Category Implicit Association Test
Perceived self image score | After 4 years of treatment
  Perceived self image score as measured through the Masculine Self Image questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Phillip, Prof, Principal Investigator — Rabin Medical Center
Locations (1):
- Schneider Children's Medical center, Petah Tikva, Israel

REFERENCES:
- [Derived] Shemesh-Iron M, Lazar L, Lebenthal Y, Nagelberg N, Tenenbaum A, Ezra R, Leffler N, Yackobovitch-Gavan M, Schoenberg-Taz M, Phillip M. Growth hormone therapy and short stature-related distress: A randomized placebo-controlled trial. Clin Endocrinol (Oxf). 2019 May;90(5):690-701. doi: 10.1111/cen.13944. Epub 2019 Mar 7. PMID 30721549